CLINICAL TRIAL: NCT05495386
Title: Investigation of Hypoglycaemia-induced EEG Changes in Participants With Type 1 Diabetes by Use of the Hyposafe H02 Device
Brief Title: Investigation of Hyposafe H02 Device in Patients With Type 1 Diabetes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawn due to company interest and development of alternative devices for epilepsy
Sponsor: UNEEG Medical A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: U010
Record Dates: First submitted 2022-05-24; First posted 2022-08-10 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hyposafe H02 Device (Experimental): Hyposafe H02 Device will be used in the study
  Interventions: Device: Hyposafe hypoglycaemia notification device (H02)

INTERVENTIONS:
Device: Hyposafe hypoglycaemia notification device (H02) — The H02 device consists of two parts:
  1. An implantable part which records the EEG signal and transmits the signal wirelessly to the external device.
  2. The external device receiving signals and storing data from the implant.
  Other Names: H02

SUMMARY:
This clinical study is designed to collect data for further development of a hypoglycaemia notification algorithm. In addition, information regarding safety will be collected and analysed.

DETAILED DESCRIPTION:
H02 is an implantable continuous EEG recorder that consists of an implant and an external device. The H02 system is based on a subcutaneous EEG measurement and acquisition of the EEG signal from the implant.

Participant will have the implantable part of H02 implanted under local anaesthesia. After a healing period, the participants will start using the external part of H02. They will wear the external part of H02 as much as possible both during daytime and night-time. The participant will use their own continuous glucose monitoring (CGM) during the study as normal practice. The participants will be exposed to insulin-induced hypoglycaemia once during the study.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Type 1 diabetes diagnosed at least five years prior to inclusion in the study
* Age 18-70 years
* Impaired awareness, i.e., defined as unaware by the Pedersen-Bjergaard scale and history of at least one severe hypoglycaemia within the preceding year
* Use of continuous glucose monitoring at study start

Exclusion Criteria:

* High risk of surgical complications
* Involved in therapies with medical devices that deliver electrical energy into the area around the implant
* Infection at the site of device implantation
* Contraindications to the local anaesthetic used during implantation and explantation
* Have cochlear implant(s)
* Subject is scheduled to undergo MRI scan, ultrasound, radiation, or electrical current induced close to the implant, within 6 months after enrolment
* Severe cardiac disease
* History of stroke/ cerebral haemorrhage and any other structural cerebral disease
* Active cancer or cancer diagnosis within the past 5 years

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
To collect electrocardiogram (EEG) data to develop a hypoglycaemia notification algorithm. | 7-8 months
  Recording of EEG characteristic hypoglycaemic related changes and EEG during normoglycemia measured as number of hours EEG data from each participant.
To collect self-measured blood glucose (SMBG) data to develop a hypoglycaemia notification algorithm. | 7-8 months
  Number SMBG measurements below 3 mmol/L glucose per participant
To collect continuous glucose monitoring (CGM) data to develop a hypoglycaemia notification algorithm. | 7-8 months
  Number of CGM values below 3 mmol/L glucose per participant

SECONDARY OUTCOMES:
To evaluate the safety of H02 in participants with type 1 diabetes. | 7-8 months
  * Number of adverse events 29 weeks after implantation (from visit 3 to visit 14)
  * Number of adverse device effects (ADEs) 29 weeks after implantation (from visit 3 to visit 14)
To evaluate the performance of H02 in participants with type 1 diabetes. | 7-8 months
  Number of device deficiencies (from visit 3 to visit 13)
To evaluate the surgeon satisfaction of H02 in participants with type 1 diabetes. | 0 and 7-8 months
  Surgeon satisfaction will be evaluated by questionnaires after the implantation at visit 3 and after explantation at visit 13 of the implantable part of Hyposafe H02 Device